CLINICAL TRIAL: NCT04035239
Title: An Open-Label Phase Ib Study to Evaluate Retinal Imaging After Short-term Use of the Balance Goggles System (BGS) in Patients With Glaucoma
Brief Title: Retinal Effects of Balance Goggles System in Glaucoma Balance Goggles System (BGS) in Patients With Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey L Goldberg, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50800
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- BGS use (Experimental): Use of BGS goggles for a 3-6 weeks period.
  Interventions: Device: BGS goggles

INTERVENTIONS:
Device: BGS goggles — BGS goggles use for 3-6 weeks

SUMMARY:
This is an open-label trial of 20 study participants with glaucoma or ocular hypertension. Participants with qualifying study eye(s) after screening and baseline evaluations will receive the Balance Goggles System. After a baseline evaluation (prior to negative pressure application through the BGS), study eyes will be treated for one hour in the clinic and be evaluated again. They will then use the BGS for the next 3-6 weeks and be evaluated again. The goal is to determine whether the intraocular pressure (IOP)-lowering effects of BGS is accompanied by changes in retinal thickness measured by optical coherence tomography (OCT), retinal vascular density measured by OCT-angiography, or retinal fluorescence measured by a fundus camera.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be medically able to undergo the testing required in the schedule of events (SOE).
2. Participant's clinical diagnosis must be consistent with glaucoma characterized by clinical evidence of progressive retinal ganglion cell dysfunction and degeneration using at least one visual field and at least one structural modality, OR with ocular hypertension with intraocular pressure above 21 mm Hg.
3. If a participant has two eyes meeting study criteria, both may be enrolled.
4. Subjects with orbital anatomy that permits a proper seal in both eyes when goggles are placed over eyes and can tolerate measurements with goggles in place
5. Participant must understand and sign the informed consent. If the participant's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the participant in its entirety.

Exclusion Criteria:

1. Subjects with a history of allergy to primary study device material (i.e., silicone)
2. Subjects with a history of any ocular disorder or condition (e.g., corneal transplant) in either eye that would likely interfere with the interpretation of the study results or compromise subject safety
3. Subjects with a prior retinal detachment, active retinal detachment, an untreated retinal detachment, unresolved cystoid macular edema, or any other fundus findings that may prevent visualization of the retina in either eye; subjects with macular degeneration are not excluded from participation in the study
4. Subjects with a history of prior penetrating glaucoma surgery (e.g. trabeculectomy, tube shunt, etc.) in either eye
5. Subjects with narrow anterior chamber angle anatomy in either eye as visualized by gonioscopy with a Shaffer angle grade of ≤ 2 in any of the four quadrants
6. Subjects with eyelid edema, festoons or excessive skin laxity in either eye
7. Subjects with conjunctival chemosis in either eye
8. Subjects with best corrected visual acuity of 20/200 or worse in either eye due to glaucoma
9. Subjects who have had intraocular surgery in the study eye within 12 weeks prior to the screening visit , or who, in the opinion of the investigator, may require any ocular surgery (e.g., cataract extraction or glaucoma procedure) in either eye during the course of the study
10. Subjects who do not wish to or cannot comply with study procedures, including home use of the study device
11. Subjects with any physical or mental condition that would, in the opinion of the investigator, increase the risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Retinal thickness | Over a 3-6 week treatment period to study completion
  Change from baseline in retinal nerve fiber layer thickness measured by optical coherence tomography imaging
Retinal vascular density | Over a 3-6 week treatment period to study completion
  Change from baseline in vessel density measured by optical coherence tomographic angiography imaging
Retinal fluorescence | Over a 3-6 week treatment period to study completion
  Change from baseline in flavoprotein fluorescence measured by fundus photography imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Byers Eye Institute at Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sun MT, Beykin G, Lee WS, Sun Y, Chang R, Nunez M, Li KZ, Knasel C, Rich C, Goldberg JL. Structural and Metabolic Imaging After Short-term Use of the Balance Goggles System in Glaucoma Patients: A Pilot Study. J Glaucoma. 2022 Aug 1;31(8):634-638. doi: 10.1097/IJG.0000000000002066. Epub 2022 Jun 13. PMID 35696700